CLINICAL TRIAL: NCT05092958
Title: MAIN-CAV: Phase III Randomized Trial of Maintenance Cabozantinib and Avelumab vs Maintenance Avelumab After First-Line Platinum-Based Chemotherapy in Patients With Metastatic Urothelial Cancer
Brief Title: Testing the Addition of the Anti-cancer Drug, Cabozantinib, to the Usual Immunotherapy Treatment, Avelumab, in Patients With Metastatic Urothelial Cancer, MAIN-CAV Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-11166; NCI-2021-11166 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A032001 (Other: Alliance for Clinical Trials in Oncology); A032001 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Bladder Urothelial Carcinoma; Advanced Renal Pelvis Urothelial Carcinoma; Advanced Ureter Urothelial Carcinoma; Advanced Urethral Urothelial Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Stage III Bladder Cancer AJCC v8; Stage III Renal Pelvis and Ureter Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Renal Pelvis and Ureter Cancer AJCC v8; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — avelumab; Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (avelumab) (Active Comparator): Patients receive avelumab IV over 60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days for 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan at screening and undergo CT or MRI and biospecimen collection throughout the trial. Patients may undergo urine sample collection as clinically indicated.
  Interventions: Drug: Avelumab; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (avelumab, cabozantinib) (Experimental): Patients receive avelumab IV over 60 minutes on days 1 and 15 of each cycle and cabozantinib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan at screening and undergo CT or MRI and biospecimen collection throughout the trial. Patients may undergo urine sample collection as clinically indicated.
  Interventions: Drug: Avelumab; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB 0010718C; MSB-0010718C; MSB0010718C
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm B (avelumab, cabozantinib)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of adding cabozantinib to avelumab versus avelumab alone in treating patients with urothelial cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cabozantinib and avelumab together may further shrink the cancer or prevent it from returning/progressing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of cabozantinib (cabozantinib S-malate) in combination with avelumab on overall survival (OS) compared to avelumab alone in patients with metastatic urothelial cancer (mUC) who did not progress during first-line platinum-based chemotherapy therapy, i.e. patients who had complete response (CR), partial response (PR) or stable disease (SD) after completion of first line platinum-based chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the effect of cabozantinib in combination with avelumab on progression-free survival (PFS) compared to avelumab alone for maintenance treatment following initial first-line treatment in patients who had a CR, PR or SD upon completion of first-line platinum-based chemotherapy.

II. To evaluate the safety and tolerability of cabozantinib in combination with avelumab in mUC compared to avelumab alone for maintenance treatment following initial first-line treatment in patients who had a CR, PR or SD upon completion of first-line platinum-based chemotherapy.

III. To evaluate activity of cabozantinib in combination with avelumab based on Response Evaluation Criteria in Solid Tumors (RECIST) compared to avelumab alone for maintenance treatment following initial first-line treatment in patients who had a CR, PR or SD upon completion of first-line platinum-based chemotherapy.

IV. Results of the primary analysis will be examined for consistency, while accounting for the stratification factors and/or covariates of baseline quality of life (QOL) and fatigue.

V. To evaluate the activity of cabozantinib in combination with avelumab compared to avelumab alone based on PD-L1 status of patients' tumors.

QUALITY OF LIFE (QOL) OBJECTIVES:

I. To compare quality-adjusted survival between patients randomized to receive cabozantinib and avelumab versus (vs.) avelumab alone using the European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L).

II. To compare patient-reported fatigue as assessed by the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue 4a from baseline through 12 months between patients randomized to receive cabozantinib and avelumab vs. avelumab alone.

III. To compare patient-reported global health status/quality of life as assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30 from baseline through 12 months between patients randomized to receive cabozantinib and avelumab vs. avelumab alone.

IV. To compare scale scores of the EORTC QLQ-Bladder Cancer Muscle-Invasive (BLM)30 (urinary symptoms, urostomy problems, catheter problems, future perspectives, abdominal bloating and flatulence, body image, sexual function) at 3, 6, 12, 18, and 24 months between patients randomized to receive cabozantinib and avelumab vs. avelumab alone.

V. To compare scale scores of the EORTC QLQ-C30 (global health status/quality of life; physical, role, emotional, cognitive, and social function; symptoms) at 3, 6, 12, 18, and 24 months between patients randomized to receive cabozantinib and avelumab vs. avelumab alone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive avelumab intravenously (IV) over 60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days for 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan at screening and undergo computed tomography (CT) or magnetic resonance imaging (MRI) and biospecimen collection throughout the trial. Patients may undergo urine sample collection as clinically indicated.

ARM B: Patients receive avelumab IV over 60 minutes on days 1 and 15 of each cycle and cabozantinib orally (PO) daily on days 1-28 of each cycle. Cycles repeat every 28 days for 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone scan at screening and undergo CT or MRI and biospecimen collection throughout the trial. Patients may undergo urine sample collection as clinically indicated.

After completion of study treatment, patients are followed every 30 days through 90 days, then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed diagnosis of advanced or metastatic urothelial cancer of the renal pelvis, ureter, bladder, or urethra (transitional cell and mixed transitional/non-transitional cell histologies except for small-cell histology), including N3 only disease prior to start of first-line platinum-based chemotherapy
* Prior first-line treatment must have consisted of 4-6 cycles of 1st-line therapy (platinum-based chemotherapy; gemcitabine-cisplatin, gemcitabine-carboplatin, methotrexate, vinblastine, doxorubicin and cisplatin [MVAC] or dose-dense [dd]MVAC)
* No more than 1 line of prior chemotherapy for metastatic or locally advanced disease (neoadjuvant or adjuvant chemotherapy will be allowed if given 12 or more months prior to registration)
* Tumor objective response of CR, PR, or SD upon completion of first line platinum-based chemotherapy by treating physician's assessment
* The last dose of first-line chemotherapy must have been received no less than 3 weeks, and no more than 10 weeks, prior to randomization in the present study
* No prior immunotherapy with IL-2, IFN-alpha, or an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects
* Women of childbearing potential must have a negative pregnancy test =< 14 days prior to registration.

  * Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Post menopause is defined as amenorrhea >= 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* No use of immunosuppressive medication within 7 days prior to randomization except:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with diabetes type I, vitiligo, psoriasis, or hypo or hyperthyroid disease not requiring immunosuppressive treatment are eligible
* None of the following:

  * Active autoimmune disease that might deteriorate when receiving the anti PD-L1 agent, avelumab.
  * No known symptomatic central nervous system (CNS) metastases. Patients with previously diagnosed CNS metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to randomization, have discontinued corticosteroid treatment for at least 2 weeks, and are neurologically stable. Baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility.
  * No major surgery within 4 weeks prior to randomization. Subjects must have complete wound healing from surgery before randomization. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
  * No palliative radiotherapy within 48 hours prior to patient randomization.
  * No hemoptysis of ≥ 0.5 teaspoon (2.5 mL) of red blood, clinically significant hematuria, hematemesis, coagulopathy, or other history of significant bleeding (eg. Pulmonary hemorrhage) within 3 months before randomization.
  * No known cavitating pulmonary lesion(s) or known endobronchial disease manifestation.
  * No administration of a live, attenuated vaccine within 30 days prior to randomization. The use of inactivated (killed) vaccines for the prevention of infectious disease is permitted. The use of COVID-19 vaccines is permitted.
  * No uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    * Cardiovascular disorders including:

      * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening.
      * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
      * The patient has a known history of corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms and confirmed by electrocardiogram (ECG) within 28 days before randomization. Note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.
      * Any history of congenital long QT syndrome.
      * Stroke, transient ischemic attack (TIA), myocardial infarction, or other symptomatic ischemic event or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism [DVT/PE]) within 6 months before randomization. Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if asymptomatic and stable at screening and treated with low molecular weight heparin (LMWH) or the direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban for at least 1 week before randomization. Non-symptomatic white matter disease in the brain is acceptable.
    * No significant gastrointestinal disorders, particularly those associated with a high risk of perforation or fistula formation including unresolved active peptic ulcer disease, cholecystitis, diverticultis, symptomatic cholangitis or appendicitis, or malabsorption syndrome within 28 days of randomization.
    * No other clinically significant disorders such as:

      * Any active infection requiring systemic treatment within 14 days before randomization. Subjects receiving oral (including prophylactic) antibiotics with no symptoms of infection at randomization are eligible.
      * Serious non-healing wound/ulcer/bone fracture within 28 days before randomization
      * History of organ or allogeneic stem cell transplant
    * No persisting toxicity related to prior therapy grade > 2 constituting a safety risk based on the investigator's judgment.
    * No diagnosis of any other malignancy within 3 years prior to randomization, except for locally curable cancers that have been adequately treated such as basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, Gleason < 7 prostate cancer on surveillance without any plans for treatment intervention (eg, surgery, radiation, or castration), or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms and no indication for treatment.
    * No concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel).

      * Allowed anticoagulants are the following:

        * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 8 g/dL
* Calculated (Calc.) creatinine clearance >= 30 mL/min using the Cockcroft-Gault equation
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN (or =< 5 x ULN for patients with liver metastases or Gilbert's disease)
* Urine protein creatinine (UPC) ratio =< 1 or 24-hour protein < 1 g
* Physicians should consider whether any of the following may render the patient inappropriate for this protocol:

  * Psychiatric illness which would prevent the patient from giving informed consent.
  * Uncontrolled medical conditions which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
  * Patients who cannot swallow oral formulations of the agent(s).

In addition:

* Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Include as applicable: Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom).
* Patients with rheumatoid arthritis and other rheumatologic arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and or steroids equivalent to < 10 mg prednisone daily, not on immunosuppressive medications and patients with positive serology are eligible. Patients with vitiligo, endocrine deficiencies including hypo or hyper thyroid disease managed with replacement, diabetes type 1 are eligible.
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the study and continue for 4 months after the last dose of study drugs, even if oral contraceptives are also used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time from randomization until death due to any cause, assessed up to 5 years
  Subgroup analyses will be done using a stratified Cox model that includes the treatment arm assignment as an explanatory variable and a separate model will be generated for each level for the subgroup of interest.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from randomization until disease progression as assessed by the treating physician using Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause, assessed up to 5 years
  A stratified Cox model will be used to compare the outcomes between the two treatment groups. The subgroup analyses will be done using a stratified Cox model that includes the treatment arm assignment as an explanatory variable and a separate model will be generated for each level for the subgroup of interest.
Tumor response | Up to 5 years
  Will be defined as a complete response or partial response (PR) as measured with Immune-Modified RECIST. Will be compared between the arms using a Mantel-Haenszel test (that accounts for the randomization stratification factors) comparing the response rates between the two treatment arms. This analysis will only include patients who had a PR or stable disease (SD) response to first-line therapy. An additional analysis will be conducted using logistic regression analysis that includes treatment arm and any baseline variables that are imbalanced between the arms as explanatory variable.
Incidence of adverse events (AE) | Up to 5 years
  Will be assessed by Common Terminology Criteria for Adverse Events 5.0. Will be summarized with frequencies and relative frequencies. The maximum grade for an AE will be recorded for each patient by treatment arm. The number (percent) of patients that experience each observed adverse event will be summarized by treatment arm. In addition, the proportion of patients that experience a grade 3+, grade 4+, and grade 5 adverse event will be summarized as the number and percent of patients by treatment arm. The primary summary will be regardless of attribution. Will also do an analogous summary for the adverse events that were deemed at least possibly related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Gupta, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (276):
- United States (272):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Baptist Health Louisville, Louisville, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Health Medical Group - Andrews Patel Hematology/Oncology East, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - University Cancer Specialists - Alcoa, Alcoa, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Valley Medical Center, Renton, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT05092958/ICF_000.pdf